CLINICAL TRIAL: NCT02774863
Title: Regional Prospective Multicenter Pilot Study: How to Collect the Expression of Psychological Suffering of Children Under Two Years ?
Brief Title: How to Collect the Expression of Psychological Suffering of Children Under Two Years?
Acronym: RESOPSYBB
Status: Terminated | Type: Observational
Why Stopped: Not enough inclusion
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0445
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Emotional Neglect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group "Maternal and Child Protection": Followed by the doctor and pediatric nurse of the Maternal and Child Protection . A child psychiatric consultation (usual care) can take place during the monitoring of this patient.
- Group "Home passages": A child psychiatric consultation is scheduled in the month following the inclusion and three home passages between the 2nd and 3rd months of follow up.
  Interventions: Other: Home passages

INTERVENTIONS:
Other: Home passages — Three home passages between the 2nd and 3rd months of follow up.
  Groups: Group "Home passages"

SUMMARY:
Emotional Neglect (NE) is a form of abuse to the child whose prevalence is high (WHO Europe). Experiencing NE, psycho-emotional development and brain child may be impacted generating psychic suffering signs may progress to severe developmental disorders. The recognition of suffering can prevent and treat these disorders.

This research promotes a multi-professional device, centered on observation, collection of expression of the baby's psychic pain (≤ 2 years) living in vulnerable families. The investigators assume that this collection requires the crossing of looks of a child psychiatrist and a repeated observation at home by a trained nurse.

The two devices described in these two groups are devices set up as part of the routine management of these patients. Usually, depending on the means of structures (human and financial), one of these devices may be preferred over another.

ELIGIBILITY:
Inclusion Criteria:

* Families say vulnerable falling M.Heaman selection criteria associated with two significant items of Q-Sort, agreeing to participate in the research project.
* Patient 24 months or less at the time of the first consultation PMI.
* Parents / legal representatives agreeing to participate in the research project.

Non inclusion Criteria:

* Serious genetic and somatic pathologies resulting deficiency, physical pain,
* Non-French speaking families.
* Families whose baby is monitored as part of the network grow together because of their prematurity.
* Minor or major Parents Trust

Ages: 1 Year to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fifty children and their families (parents / guardians) will be included in the research in the department of Loire-Atlantique, coming visit to the Mother and Child Protection within the first two years of their child.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the sensitivity of the Global Printing-scale gravity relative to the Development Quotient (reference) between the 2 supported (Group A versus Group B). | up to three months
  Development Quotient level will be measured by Brunet Lezine R. This questionnaire provides an objective measure of the impact of mental suffering. It will be measured by psychomotor between the 3rd and 4th month follow up.
  A child with a score of QD lower or equal 85 is considered a child with developmental impairment.
  - Clinical Global Impression Severity Scale suitable for measuring the assessment of mental suffering of children less than two years is considered an indicator of the intensity of suffering. This will be assessed by a nurse between the 3rd and 4th months of follow up.
  A child with a CGI-severity score between 1 and 4 inclusive shall be considered a child with developmental impairment.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Medical-social Center Dalby Millet, Nantes
  - Medical-Social center Bellevue, Nantes
  - Medical-social center Pilotière, Nantes
  - Medical-Social center Port Boyer, Nantes
  - Medical-social St-Etienne de Montluc, Saint-Étienne-de-Montluc
  - Medical-social Saint-Servan, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No